CLINICAL TRIAL: NCT01831375
Title: Health Care Partners in Cancer Prevention and Care Among Aged
Brief Title: Cancer Prevention and Care Among Aged
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Eva Kahana, Ph.D., Distinguished University Progessor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA098966-07 (NIH)
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Speak Up (Experimental): Participants will learn how to speak up to their medical doctors for improving their medical care.
  Interventions: Behavioral: Speak Up
- Get Connected (Other): Attention control group
  Interventions: Behavioral: Get connected

INTERVENTIONS:
Behavioral: Speak Up — Intervention group_treatment group
  Other Names: The Involved Elders Project
  Arms: Speak Up
Behavioral: Get connected — Participants will learn to be connected with social resources in the community.
  Arms: Get Connected

SUMMARY:
This research represents a pioneering effort to design a brief, cost effective and readily transportable program that will enable disadvantaged elders to become more effective participants in their health care.

The intervention is expected to result in trained elders becoming more knowledgeable health care partners. Trained patients will be prepared for appointments and will engage their primary care physicians in active dialogue regarding cancer prevention and screening.

Based on self-advocacy, these patients are expected to receive better preventive care and report greater satisfaction with care. Program participation can subsequently contribute to general health improvements and minimize health disparities.

DETAILED DESCRIPTION:
In a randomized controlled trial (RCT) with 400 older adults, the investigators will assess the efficacy of the "Speak Up" intervention (N=200) relative to an attention control group "Connect" program (N=200), aimed at enhancing social and civic engagement. Participants will now obtain resource materials that include decision aids and diary logs to bring to visits with doctors. The investigators will implement "Speak Up" and "Connect" programs in two unique study populations: 1) participants in the ongoing NCI study and 2) older adults attending senior center programs sponsored by Area Agencies on Aging (AAAs). Participants will be assessed prior to the intervention and 2 month, and 12 months post intervention. The investigators will have an observation window of 12 months to determine whether and when the older adult obtained screening. The selection of a shorter follow-up time frame will help reduce attrition.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Over the age of 65 from Area Agencies of Aging who are interested in participating

Exclusion Criteria:

* No exclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 697 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Perception of Physician Quality Scale | one year
  Perception of Physician Quality Scale(Lee & Kasper, 1998) will be used to measure patient satisfaction with physician care (p. 21). Questions include satisfaction with physician visits and satisfaction with physician knowledge of respondent's medical problems. This scale has been utilized with elderly populations (e.g. Burton et al. 2002) and has been found to be a valid and reliable (Cronbach's alpha greater than .8) measure of patient satisfaction (Lee & Kasper, 1998).

SECONDARY OUTCOMES:
Cancer Screening Recommendations | one year
  Physicians would make more recommendations for cancer prevention and screening

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kahana, Ph.D., Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States